CLINICAL TRIAL: NCT02539810
Title: Optimum and Stepped Care Standardised Antihypertensive Treatment With or Without Renal Artery Stenting in Patients With Documented Resistant Hypertension and Atherosclerotic Renal Artery Stenosis. ANDORRA TRIAL
Brief Title: Renal Artery Stenting in Patients With Documented Resistant Hypertension and Atherosclerotic Renal Artery Stenosis (ANDORRA)
Acronym: ANDORRA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P140914; P140914 (Other: DRCD)
Record Dates: First submitted 2015-07-28; First posted 2015-09-03 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Hypertension; Hypertension Resistant to Conventional Therapy; Angiographically Proven Grade III Unilateral or Bilateral Atherosclerotic Renal Artery Stenosis (ARAS) Greater Than or Equal to 60 Percent
MeSH Terms: conditions — Hypertension; Hypertension Resistant to Conventional Therapy | interventions — Stents; Antihypertensive Agents; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal artery stenting (Experimental): Renal artery angioplasty plus stenting and standardized and optimized medication regimen.
  Patients are treated with renal artery stenting plus a standardized optimal medical treatment, including the antihypertensive treatment which is adapted every month starting two month after randomization on the basis of home BP monitoring results at follow-up visits.
  Interventions: Device: Renal artery Angioplasty plus stenting.; Drug: Anti hypertensive, statin and antiplatelet medication.
- standardized and optimized medication regimen (Active Comparator): Patients are treated with a standardized optimal medical treatment including the antihypertensive treatment which is adapted every month starting two month after randomization on the basis of home BP monitoring results at follow-up visits.
  Interventions: Drug: Anti hypertensive, statin and antiplatelet medication.

INTERVENTIONS:
Device: Renal artery Angioplasty plus stenting. — renal artery stenting
  Other Names: RA Stent
  Arms: Renal artery stenting
Drug: Anti hypertensive, statin and antiplatelet medication. — Slow release indapamide 1.5 mg/d (or furosemide 40 mg/d if eGFR is < 30 mL/min/1.73m²) + irbesartan 300 mg/d + amlodipine 10 mg/d + aspirin 75 mg/d (or clopidogrel 75 mg/d in case of allergy or gastrointestinal intolerance to aspirin) + atorvastatin 20 mg/d. After randomization, bisoprolol 10 mg/d, prazosin 5 mg/d, and rilmenidine 1 mg/d and spironolactone 12.5 to 25 mg/d, will be sequentially added from months two to five in both groups if home blood pressure remains more than or equal to 135/85 mm Hg.
  Other Names: SOMT

SUMMARY:
The ANDORRA study is a, multicenter, prospective, open, randomized, controlled blinded endpoint trial (PROBE) comparing two treatment strategies (renal artery stenting + standardized and optimized medical treatment [SOMT] versus SOMT alone) of 12 months duration in patients with confirmed resistant hypertension (RH) and angiographically proven grade III unilateral or bilateral atherosclerotic renal artery stenosis (ARAS) ≥ 60%.

DETAILED DESCRIPTION:
All eligible patients diagnosed with RH on office BP measurements and unilateral or bilateral ARAS ≥60% on a non-invasive test (CT-angiogram or MR-angiogram) will receive a standardized optimized triple antihypertensive treatment for 4 weeks. After 4 weeks, patients with confirmed RH by ABPM (daytime ABPM ≥ 135 or 85 mmHg) and no clinically significant increase in plasma creatinine from baseline (< 30%) will undergo a renal angiogram to confirm the degree of ARAS ≥60% in diameter.

Immediately after the renal angiography, all patients will undergo flow fractional reserve (FFR) measurements. Once FFR measurements have been done and all criteria are met, patients will be randomized in the angiography room to either renal artery stenting + SOMT (stenting group) versus SOMT (control group) whatever the results of the FFR in a 1:1 ratio. Both groups will continue the SOMT during follow-up.

The SOMT will be prescribed from the inclusion visit until the 6 month-visit after randomization. After randomization, the antihypertensive treatment will be adapted according to the results of home BP (HBP) at monthly visits starting 2 months after randomization. After the 6-month visit, the antihypertensive treatment adaptation will be left at the discretion of the physician in charge of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 80 Years
* Men or women
* Supine office BP ≥ 140 and/or 90 mmHg at screening despite a stable medication regimen including full tolerated doses of 3 or more anti-hypertensive treatments of different classes, including a diuretic.
* Unilateral or bilateral ARAS of a main renal artery ≥60% diagnosed by renal CT- angiogram (or MR-angiogram if there is a contraindication to perform CT) performed in the year before
* One or two functional kidney(s) ≥ 70 mm in pole-to-pole length
* eGFR ≥ 20 ml/min/1.73 m² (MDRD formula)
* Signed informed consent
* Social insurance coverage

Inclusion criteria for the renal angiogram procedure:

- RH confirmed by daytime ABPM ≥ 135 or 85 mmHg after 1 month treatment with SOMT at Visit V1.

Inclusion criteria for the randomization:

* Unilateral or bilateral ARAS of a main renal artery ≥ 60% confirmed on renal angiogram by Quantitative Vascular Analysis (QVA)
* Increase in plasma creatinine < 30% after 4-week SOMT

Exclusion Criteria:

* Fibromuscular dysplasia of renal artery or other non-atherosclerotic renal artery stenosis
* Other secondary form of hypertension excluded on the basis of a clinical, hormonological and/or imaging work-up
* Restenosis after a previous renal angioplasty or stenting
* Only a stenosis of an accessory renal artery supplying <1/2 of the ipsilateral renal parenchyma
* Additional indication of ARAS stenting (Malignant hypertension, ≥ 30% increase in plasma creatinine after renin angiotensin system (RAS) blocker or after RAS blocker and diuretic administration, flash pulmonary edema)
* Kidney pole-to-pole length < 70 mm
* Vascular disease precluding access for stenting
* Abrupt vessel closure or dissection after diagnostic angiography
* Contraindication to renal artery stenting according the notice for use of the stents
* eGFR < 20 ml/min/1.73 m² (MDRD)
* History of transient ischemic accident (TIA) or cerebrovascular accident (CVA) during the 3 months prior to visit 1
* History of acute heart failure or heart failure (NYHA class III-IV) within the 3 months prior to visit 1
* History of myocardial infarction, unstable angina, coronary bypass or percutaneous coronary angioplasty during the 3 months prior to visit 1
* Abdominal aortic aneurysm with indication for surgery or EVAR (Endovascular Aneurysm Repair)
* Known history of cholesterol embolism
* Brachial circumference of ≥ 42 cm
* Severe contrast media allergy, not amenable to pre-treatment
* Allergy to aspirin or clopidogrel
* Atrial fibrillation
* Comorbid condition causing life expectancy ≤ 3 years
* Unlikely to co-operate in the study and/or poor compliance anticipated by the investigator
* Participant not affiliated to the French social security
* Pregnancy or breastfeeding
* Guardianship for incapacity

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Mean change in diurnal systolic blood pressure assessed by ambulatory BP monitoring (ABPM) | Baseline to 6 months

SECONDARY OUTCOMES:
Adverse events of renal artery stenting | Baseline to 12 months
Change in average 24-hour and nighttime Systolic Blood Pressure by ABPM | Baseline to 12 months
Change in average 24-hour, daytime and nighttime diastolic Blood Pressure by ABPM | Baseline to 12 months
Change in Systolic/diastolic Blood Pressure by home blood pressure monitoring | Baseline to 12 months
Change in office Systolic/diastolic Blood Pressure | Baseline to 12 months
Antihypertensive medication score | Baseline to 12 months
Detection of the drugs in urine by LC-MS/MS | Baseline to 12 months
Renal artery restenosis in patients of the stenting group assessed by duplex ultrasound and/or renal CTA | Baseline to 12 months
Adverse cardiovascular (CV) events | Baseline to 12 months
Change in plasma creatinine and eGFR | Baseline to 12 months
Clinical renal events: renal death, progressive renal insufficiency (i.e. need for dialysis), need for permanent renal replacement therapy, need of target vessel stenting in the SOMT group (number of crossovers) | Baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michel AZIZI, Principal Investigator — HEGP - APHP
Locations (15):
- France (15):
  - Hopital Pasteur, Nice, Alpes-Maritimes
  - Hopital Saint Andre - CHU Bordeaux, Bordeaux, Gironde
  - Hopital Rangueil - CHU Toulouse, Toulouse, Haute-Garonne
  - Hopital Lapeyronie - CHU Montpellier, Montpellier, Herault
  - Hopital Arthur Gardiner, Dinard, Ille-et-Vilaine
  - Hopital Pontchaillou - CHU Rennes, Rennes, Ille-et-Vilaine
  - Groupe Hospitalier Mutualiste, Grenoble, Isere
  - Hopital Michallon - CHU Grenoble, La Tronche, Isere
  - Institut Lorrain du Cœur et des Vaisseaux Louis Mathieu, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Hopital de Brabois, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Hopital Cardiologique - CHRU Lille, Lille, Nord
  - CHU Clermont-Ferrand, Clermont-Ferrand, Puy-de-Dome
  - Hopital de la Croix-Rousse - CHU Lyon, Lyon, Rhone
  - Hopital de la Pitie Salpetriere, Paris
  - Hopital Europeen Georges Pompidou (HEGP), Paris